CLINICAL TRIAL: NCT07208279
Title: Effects of Dietary Supplement Intervention on Cognitive Function and Psychological Well-Being
Brief Title: Cognitive Vitality Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Judith Klein-Seetharaman, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022585
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Aging; Healthy Aging; Cognition; Memory; Brain

STUDY DESIGN:
Intervention Model Description: Simple random convenience sampling procedures will be used to divide the sample (n = 16) into a control group and an active group (n = 8, respectively). The RAND function in Microsoft Excel will be used as a cost-effective tool to generate a random sample and numerical identification numbers will be assigned to each participant to protect personal information.
  The active intervention group will be asked to consume 1 packet of Axolt dissolved in about 16 oz of water once a day for 45 days. The control group will be asked to consume 1 packet of Bolero flavored water mix hydration enhancement also in about 16 oz of water once a day for 45 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axolt Brain Supplement (Experimental): The active intervention group will be asked to consume 1 packet of Axolt dissolved in about 16 oz of water once a day for 45 days.
  Interventions: Dietary Supplement: Axolt Brain Supplement
- Bolero - Flavored Drink Placebo (Placebo Comparator): The control group will be asked to consume 1 packet of Bolero flavored water mix hydration enhancement also in about 16 oz of water once a day for 45 days.
  Interventions: Dietary Supplement: Bolero - Flavored Drink Placebo

INTERVENTIONS:
Dietary Supplement: Axolt Brain Supplement — https://axoltbrain.com/ Axolt is a brain health supplement. It includes native ingredients, formulated to help the brain perform at its best.
  Arms: Axolt Brain Supplement
Dietary Supplement: Bolero - Flavored Drink Placebo — The control group will be asked to consume 1 packet of Bolero flavored water mix hydration enhancement also in about 16 oz of water once a day for 45 days.
  Arms: Bolero - Flavored Drink Placebo

SUMMARY:
This study's purpose is to evaluate the effects of a dietary supplement on cognitive function and psychological well-being in community-dwelling older adults aged 55+. The study involves taking a commercially available dietary supplement daily for 45 days. A 45-minute assessment will be conducted at the beginning and again at the end of the study.

DETAILED DESCRIPTION:
The primary aim of this randomized, single-site pilot study is to evaluate the effects of the oral liquid dietary supplement Axolt (https://axoltbrain.com) on cognitive function in adults aged 55 and older without cognitive impairment, compared to a control group taking a commercially available, hydration powdered drink flavoring, Bolero (https://bolerousa.net) daily for 45 days. The secondary aim is to assess changes in mood and psychological well-being with supplement intake. The study will use validated, low-risk cognitive measures at baseline and at the end of the study to measure change over time. 20 individuals age 55 years and older will be recruited. Sample size for enrollment: (n =8) for the active group and (n=8) in the control group (16 total), accounting for an anticipated 20% drop out rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 years and older
* Live independently,
* Self-report as healthy
* Adequate vision
* Fluent in English
* No history of mild cognitive impairment
* Currently not taking dietary supplements with the same active ingredients in Axolt or naturally flavored water
* A Montreal Cognitive Assessment [12] (MOCA) score ≥ 24
* Able to provide written informed consent, and medical clearance to participate.

Exclusion Criteria:

* Previous participation in a cognitive dietary supplement study in the last 12 months
* A score of < 24 on the Montreal Cognitive Assessment (MoCA) as a potential risk for obtaining informed consent
* History of seizures
* Epilepsy
* Parkinson's disease
* History of severe head trauma
* Uncontrolled hypertension
* On psychoactive medications
* Substance abuse
* Unwilling or unable to discontinue current dietary supplements with similar ingredients
* Planned surgery during the study period
* Medications known to interact with active ingredients with Axolt
* Minors and prisoners will be excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Digit Span Forward | From enrollment to the end of treatment at 45 days.
  Digit Span Forward measures short-term memory (5 min.) Score: Min = 2, Max = 8 *Higher score means better outcome
RAVLT Learning | From enrollment to the end of treatment at 45 days.
  Rey Auditory Verbal Learning Test (RAVLT) Learning assesses short-term memory (10 min).
  Score: Min = 0, Max = 105 *Higher score means better outcome
Digit Span Backward | From enrollment to the end of treatment at 45 days.
  Digit Span Backward measures working memory (5 min.). Score: Min = 2, Max = 8 *Higher score means better outcome
Symbol Digit Modalities Test (SDMT) | From enrollment to the end of treatment at 45 days.
  Symbol Digit Modalities Test (SDMT) measures perceptual speed (5 min.). Score: Min = 0, Max = 120 *Higher score means better outcome
RAVLT Recall | From enrollment to the end of treatment at 45 days.
  Rey Auditory Verbal Learning Test (RAVLT) Recall measures long-term memory (5 min.). Score: Min = 0, Max = 15 *Higher score means better outcome
Brain Fog Questionnaire | From enrollment to the end of treatment at 45 days.
  Brain Fog Questionnaire allows entry of self-reported cognitive difficulties (5 min.). Score: Min = 0, Max = 10 *Lower score means better outcome
PHQ-9 | From enrollment to the end of treatment at 45 days.
  The Patient Health Questionnaire (PHQ-9) records depressive symptoms (5 min.). Score: Min = 0, Max = 27 *Lower score means better outcome
GAD-7 | From enrollment to the end of treatment at 45 days.
  Generalized Anxiety Disorder 7-item Questionnaire (GAD-7) quantifies anxiety (5 min.). Score: Min = 0, Max = 21 *Lower score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Judith Klein-Seetharaman, PhD, Principal Investigator — Arizona State University
Locations (1):
- Community, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary outcomes will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available after all data have been collected, entered into the REDCap database, data cleaning procedures have been completed, and the primary articles have been published. Data will be available on or before 1/1/2028 and will remain available for a minimum of 3 years.
Access Criteria: The Arizona State University Research Data Repository can be accessed freely by investigators. This data repository has supporting information about the protocol and contact information for the investigative team.
URL: https://dataverse.asu.edu/